CLINICAL TRIAL: NCT00622206
Title: Pharmacokinetics of Low Dose Ritonavir in Thai Patients on a Saquinavir 1500 mg Based HAART Regimen
Brief Title: Pharmacokinetics of Low Dose Ritonavir
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 083; IRB#188/50
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: Pharmacokinetics; ritonavir; saquinavir; safety and toxicity; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Twenty HIV-infected volunteers on stable doses of SQV/RTV 1500/100 mg OD for at least 3 months with an NRTI backbone and undetectable viral load will participate. After collecting samples for a full PK curve subjects will be switched to SQV/RTV 1500 /50 mg OD + 2NRTIs for 1 week before repeating the PK assessment. Blood samples will be drawn at T 0, 1, 2, 4, 6, 8, 10, 12 and 24 hours post ingestion. Consecutively to the assessment, subjects will return to SQV/RTV 1500/100 mg OD dosage.
  Interventions: Drug: ritonavir and saquinavir

INTERVENTIONS:
Drug: ritonavir and saquinavir — saquinavir/ritonavir 1500/100 mg or 1500/50 mg Twenty HIV-infected volunteers on stable doses of SQV/RTV 1500/100 mg OD for at least 3 months with an NRTI backbone and undetectable viral load will participate. After collecting samples for a full PK curve subjects will be switched to SQV/RTV 1500 /50 mg OD + 2NRTIs for 1 week before repeating the PK assessment. Blood samples will be drawn at T 0, 1, 2, 4, 6, 8, 10, 12 and 24 hours post ingestion. Consecutively to the assessment, subjects will return to SQV/RTV 1500/100 mg OD dosage.

SUMMARY:
Compare the Pharmacokinetics of ritonavir and saquinavir(using either Saquinavir /Ritonavir 1500/100 mg or 1500/50 mg) Evaluate short term tolerability, safety and toxicity Evaluate if there is any relation between RTV concentration levels and boosting effect

DETAILED DESCRIPTION:
This study will focus on the combination of Saquinavir (SQV) and RTV. Firstly, this is because SQV is widely used in Thailand and has shown to be an adequate first and second line antiretroviral agent. Secondly, reduced dose of SQV (1600 mg OD) has proven to generate adequate efficacy and good pharmacokinetic parameters in the Thai population[5, 6]. Now 500 mg tablets of SQV are becoming more and more available, therefore a 1500 mg OD dose will be of more interest for our study. A TDM comparison study between SQV 1600 OD mg and SQV1500 mg OD has been done (Ananworanich et al, unpublished data) and did not show any difference in terms of drug concentrations . The efficacy of this regimen has shown to be adequate as described in the STACCATO cohort[7]. So we consider it safe to use the SQV 1500 mg OD in our study.

It is not clear what RTV concentrations are necessary to obtain good levels for SQV. In the study of Autar et al [5] no relation between RTV levels and boosting effect was described. Besides that it might well be that even the boosting levels of RTV contribute to the toxicity of the antiretroviral treatment.For instance, a study performed in healthy volunteers on RTV 100 mg BID monotherapy, showed a significant increase in total cholesterol, low-density lipoprotein (LDL) cholesterol and triglycerides and a marked reduction of high-density lipoprotein (HDL)[8]. This last finding was confirmed in the study of Boyd et al (submitted) in Thai HIV-infected patients.

Preliminary data from HIVNAT 019 [9] suggests that lower boosting dosage still give adequate levels of the other PIs. In this open label 4 arm study one arm contains Lopinavir/Ritonavir 266/66 mg bid together with SQV 600 mg bid. Despite the dose reduction in all PIs, adequate PK levels were obtained. Two arms (23 patients) in this study used normal dose of RTV (100 mg bid) in combination with Lopinavir and Saquinavir. Five of them had maximal concentrations (Cmax) above the therapeutic level RTV (>2.1 mg/l). This finding is supported by clinical experience.

Therefore, looking into lower doses of RTV in the Thai population is of great interest A liquid formulation for RTV 50 mg will be used, as a capsule is not available yet. The liquid formulation has the same bioequivalence as the capsule and was used extensively during the time of manufactory problems of the Norvir capsule. Because of the bad taste of this formulation PK samples will be collected after one week, thereafter patients can return to their old regimen. A dose reduction of RTV can be of great importance for the Thai population as it prevents unnecessary toxicity and costs. If this PK study turns out to be adequate, an efficacy study can be performed and the boosting of other commonly used PI's, like IDV and Lopinavir, can be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Documented positive test for HIV-1 infection
* HIV RNA viral load 50 < copies for at least 3 months
* Written informed consent
* On a Saquinavir 1500 mg based HAART regimen for at least 3 months

Exclusion Criteria:

* Pregnant or lactating
* Use of concomitant medication that may interfere with the pharmacokinetics of saquinavir/ritonavir
* Inability to understand the nature and extent of the study and the procedures required
* ALT/ AST more than 5x upper limit
* Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To compare the Pharmacokinetics od ritonavir and saquinavir in Thai HIV-1 infected subjects using either Saquinavir /Ritonavir 1500/100 mg or 1500/50 mg | 6 months and 1 week

SECONDARY OUTCOMES:
Evaluate short term tolerability, safety and toxicity of this treatment strategy Evaluate if there is any relation between RTV concentration levels and boosting effect | 6 months and 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Avihingsanon A, van der Lugt J, Kerr SJ, Gorowara M, Chanmano S, Ohata P, Lange J, Cooper DA, Phanuphak P, Burger DM, Ruxrungtham K. A low dose of ritonavir-boosted atazanavir provides adequate pharmacokinetic parameters in HIV-1-infected Thai adults. Clin Pharmacol Ther. 2009 Apr;85(4):402-8. doi: 10.1038/clpt.2008.244. Epub 2008 Dec 31. PMID 19118378
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org